CLINICAL TRIAL: NCT04424797
Title: Prone Positioning on Admission for Hospitalized COVID-19 Pneumonia Protocol
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Poudre Valley Health System (Other)
Responsible Party: Principal Investigator, Lucie Uncapher, Investigator, Poudre Valley Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-6034
Record Dates: First submitted 2020-06-05; First posted 2020-06-11 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Prone Position

STUDY DESIGN:
Intervention Model Description: Prone vs. Supine positioning
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prone Positioning (Experimental): Prone positioning
  Interventions: Other: Prone Positioning
- Supine Positioning (Other): Supine Positioning
  Interventions: Other: Supine Positioning

INTERVENTIONS:
Other: Prone Positioning — Intervention is patient in prone positioning
  Arms: Prone Positioning
Other: Supine Positioning — Intervention is patient in supine positioning
  Arms: Supine Positioning

SUMMARY:
A pilot study to investigate the effects of the prone positioning (PP) on hospital patients diagnosed with COVID-19 pneumonia.

Investigators that early self-proning may prevent intubation and improve mortality in patients with Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-COV-2).

Up to 100 participants with a primary diagnosis of confirmed COVID-19 pneumonia will be enrolled to the study.

All participants will be screened and those that meet inclusion and exclusion criteria will be enrolled to one of two groups: one with prone positioning (on the belly) and the other with standard supine positioning (on the back). The patient and nursing staff will monitor times spent in various positions.

Outcome measures include incidence of intubation, max oxygen requirements, length of hospital stay, ventilator-free days, worsening of oxygenation saturation, and mortality.

DETAILED DESCRIPTION:
In hypoxic respiratory failure, placing patients in the prone position improves ventilation to perfusion matching, alveolar recruitment, and alveolar to arterial oxygen gradients. Specifically, in Acute Respiratory Distress Syndrome ARDS, proning intubated patients improves overall mortality. With the emergence of SARS-COV-2, hospitals around the world have seen a marked increase in patients with acute hypoxic respiratory failure and ARDS. This surge in cases has prompted a search for more effective strategies to reduce intubation and improve patient morbidity and mortality. One such strategy is that of voluntary proning, in which awake patients are instructed to prone themselves (Early PP With High Flow Nasal Cannula (HFNC) Versus HFNC in COVID-19 Induced Moderate to Severe ARDS) (COVID-19 smArtphone-based Trial of Non-ICU Admission Prone Positioning (CATNAP)).

This trial proposes a voluntary proning strategy in patients admitted to the hospital, not yet requiring mechanical ventilation. Given the clear evidence that proning improves outcomes in ARDS, investigators hypothesize that early, voluntary self-proning may prevent intubation and improve mortality in patients with SARS-COV-2.

Methods

This is a pilot study of up to 100 participants at UCHealth facilities.

Patients will be assessed if they can self prone safely and be assessed against inclusion and exclusion criteria within 12 hours of admission and randomized to either prone or supine positioning. Baseline labs will be measured and all participants will be monitored continuously via pulse oximetry.

The Standard Supine Control Group will utilize standard oxygen (O2) device in supine position at approximately 30-60 degrees to target peripheral capillary oxygen saturation (SpO2) >90% and the participant or nurse will document time in non-supine position.

The Prone Experimental Group will position patient in approximately 15-degree reverse trendelenburg and prone using pillows for comfort. The participant will be asked to rotate to prone positioning every 2 hours while awake and encourage to sleep prone overnight as possible with a goal of 10-12 hours daily. Patient to log all time prone.

Treatment Failure may occur and termination of Intermittent Prone Positioning will occur. This is defined as respiratory distress or a decrease in O2 saturations <90% for more than 2 minutes as determined by bedside nursing or per virtual pulse oximetry monitoring notifications during the study on two consecutive occasions. The participant will be returned to supine positioning and follow standard supine oxygenation. The participant can be re-challenged in the prone position after the participant stabilizes for 2 hours. The participant can also choose to stop proning and would be considered a treatment failures.

Statistical Analysis and Sample Size In New York City the intubation rate has been reported at 1/3 of COVID-19 positive patients admitted to the hospital. The table below shows the sample size needed for a binomial outcome of intubation when 50% of the sample is randomized to Prone Positioning (PP):

Alpha 0.05 0.05 0.05 0.05 Beta 0.80 0.80 0.80 0.80 Probability of intubation with PP 0.05 0.10 0.15 0.20 Probability of intubation 0.33 0.33 0.33 0.33 Proportion receiving PP 0.50 0.50 0.50 0.50 Sample size 33 39 56 97

Expecting a 13% decrease in intubations with the prone position, investigators will use a sample size of N = 100 (50 per group) in order to have 80% power with a two-sided alpha = 0.05 for logistic regression. ANCOVA will be used to evaluate continuous, secondary variables in order to adjust for covariates. The study is powered for the primary outcome of intubation or no intubation. No adjustments will be made for the secondary endpoints.

The investigators and statistician will validate the data and the study will be subject to institutional quality assurance reviews.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the hospital floor with primary diagnosis of confirmed COVID-19 pneumonia and respiratory failure requiring greater than or equal to 2 Liters(L) Nasal Cannula (NC) to maintain SpO2>90%
* Ability to independently change positions in bed
* Able to tolerate prone positioning
* Age greater than 18

Exclusion Criteria:

* ICU admission on arrival
* Respiratory distress requiring immediate intubation

  * Respiratory Rate(RR)>35/min, accessory respiratory muscle use (ex. speaking in short sentences), signs of respiratory muscle fatigue, altered mental status, or inability to protect airway
* Chest or facial trauma, pneumothorax or other contraindication to prone positioning (i.e., spinal instability, recent abdominal surgery, pregnancy, etc)
* Hemodynamically unstable

  * Heart Rate (HR)>120 bpm, Systolic Blood Pressure (SBP)<90 mmHg, Mean Arterial Pressure (MAP)<65 mmHg or requirement for vasopressor
* Nausea and vomiting
* Pregnancy
* Refusal or inability to tolerate initial prone positioning due to comfort

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-07-13 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of intubation | Through study completion, an average of 6 days
  Incidence of intubation

SECONDARY OUTCOMES:
Maximum oxygen requirement | Through study completion, an average of 6 days
  Measure of maximum oxygen requirements
Length of Stay | Through study completion, an average of 6 days
  Measured in days of hospitalization
Ventilator-free days | Through study completion, an average of 6 days
  Measured in days not on a ventilator
Treatment failure of prone positioning due to worsening SpO2 status while prone | Through study completion, an average of 6 days
  Whether or not the participant met treatment failure descriptions
Mortality | Through study completion, an average of 6 days
  Whether or not the participant died while hospitalized

CONTACTS AND LOCATIONS:
Overall Officials: Lucie Uncapher, Principal Investigator — University of Colorado Health
Locations (3):
- United States (3):
  - UCHealth Poudre Valley Hospital, Fort Collins, Colorado
  - UCHealth Greeley Hospital, Greeley, Colorado
  - UCHealth Medical Center of the Rockies, Loveland, Colorado

IPD SHARING:
Plan to Share IPD: No